CLINICAL TRIAL: NCT06309433
Title: Assessment of Bone Mineral Density at the Interface With the Femoral and Tibial Components in Patients Undergoing Total Knee Prosthesis of Different Design and Material
Brief Title: Assessment of Periprosthetic Bone Mineral Density in Patients Undergoing Total Knee Prosthesis of Different Design
Acronym: DXA-TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DXA-TKA
Record Dates: First submitted 2024-01-13; First posted 2024-03-13 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Periprosthetic Osteolysis
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS TKA (Active Comparator): Patients with Posterior stabilized Total knee replacement
  Interventions: Diagnostic Test: dual energy x-ray absorptiometry
- CR TKA (Active Comparator): Patients with cruciate retaining Total knee replacement
  Interventions: Diagnostic Test: dual energy x-ray absorptiometry

INTERVENTIONS:
Diagnostic Test: dual energy x-ray absorptiometry — Patient will undergo periodic (6-12-24m) dexa scans on the periprosthetic bone

SUMMARY:
compare changes in BMD via DXA at the level of the femoral and tibial periprosthetic bone between two groups of patients undergoing cemented TKA of different design (posterior stabilization vs posterior cruciate preservation) with proms at a 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 45 years
2. Patients who are candidates for primary cemented total knee replacement based on physical examination and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

to. Primary or secondary osteoarthritis b. Collagen disorders and/or avascular necrosis of the femoral condyle c. Moderate valgus, varus or flexion deformities (HKA within ±10°, flexion contracture <10°) 3. Patients consenting and able to complete planned study procedures and follow-up assessments 4. Patients informed about the nature of the study who signed the "informed consent" approved by the ethics committee.

Exclusion Criteria:

1. Patients aged < 45 years;
2. Patients who have already undergone hip or knee arthroplasty ankle, previous osteotomy, with severe axial deformities or suffering from rheumatoid arthritis, diabetes or neuromuscular diseases. In this way, homogeneity of the investigated cohort will be guaranteed;
3. Pregnant women. -

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Periprosthetic bone mineral density measurement | at baseline (day 0)
  measurement of periprosthetic bone mineral density using dual-energy x-ray absorptiometry
Periprosthetic bone mineral density measurement | 6 months
  measurement of periprosthetic bone mineral density using dual-energy x-ray absorptiometry
Periprosthetic bone mineral density measurement | 12 months
  measurement of periprosthetic bone mineral density using dual-energy x-ray absorptiometry
Periprosthetic bone mineral density measurement | 24 months
  measurement of periprosthetic bone mineral density using dual-energy x-ray absorptiometry

SECONDARY OUTCOMES:
Knee Society Score | at baseline (day 0)
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Knee Society Score | 6 months
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Knee Society Score | 12 months
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Knee Society Score | 24 months
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Western Ontario and McMaster Universities Arthritis Index | at baseline (day 0)
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Western Ontario and McMaster Universities Arthritis Index | 6 months
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Western Ontario and McMaster Universities Arthritis Index | 12 months
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Western Ontario and McMaster Universities Arthritis Index | 24 months
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Knee injury and Osteoarthritis Outcome Score | at baseline, (day 0)
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living, Function in Sport and Recreation, and knee-related Quality of Life . the score goes from 0 to 100
Knee injury and Osteoarthritis Outcome Score | 6 months
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living , Function in Sport and Recreation , and knee-related Quality of Life . the score goes from 0 to 100
Knee injury and Osteoarthritis Outcome Score | 12 months
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living , Function in Sport and Recreation , and knee-related Quality of Life . the score goes from 0 to 100
Knee injury and Osteoarthritis Outcome Score | 24 months
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living , Function in Sport and Recreation , and knee-related Quality of Life . the score goes from 0 to 100
36-Item Short Form Health Survey | at baseline (day 0)
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
36-Item Short Form Health Survey | 6 months
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
36-Item Short Form Health Survey | 12 months
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
36-Item Short Form Health Survey | 24 months
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Stefano Zaffagnini, Bologna, Italia
  - Istituto ortoepdico rizzoli, Bologna

IPD SHARING:
Plan to Share IPD: No